CLINICAL TRIAL: NCT02483000
Title: Evaluation of Pretargeted Anti-CD20 Radioimmunotherapy Combined With BEAM Chemotherapy and Autologous Stem Cell Transplantation for High-Risk B-Cell Malignancies
Brief Title: Anti-CD20 Radioimmunotherapy Before Chemotherapy and Stem Cell Transplant in Treating Patients With High-Risk B-Cell Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed early due to lack of funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9189; NCI-2015-00299 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9189 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA044991 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2015-06-23; First posted 2015-06-26 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-09

CONDITIONS: Burkitt Lymphoma; CD20-Positive Neoplastic Cells Present; Diffuse Large B-Cell Lymphoma; Indolent Non-Hodgkin Lymphoma; Mantle Cell Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Refractory Mature B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Indium; Melphalan; Peripheral Blood Stem Cell Transplantation; DOTA-biotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PRIT) (Experimental): B9E9-FP INFUSION: Patients receive B9E9-fusion protein IV over a minimum of 2 hours on day -17.
  CLEARING AGENT INFUSION: Patients receive clearing agent IV over a minimum of 30 minutes on day -15.
  RADIOBIOTIN INFUSION: Patients receive indium In 111-DOTA-biotin IV and yttrium Y 90 DOTA-biotin IV over 2-5 minutes on day -14.
  BEAM CHEMOTHERAPY: Patients receive BEAM chemotherapy comprising carmustine IV over 3 hours on day -7; etoposide IV over 2 hours BID and cytarabine IV over 4 hours BID on days -6 to -3; and melphalan IV over 30 minutes on day -2.
  STEM CELL INFUSION: Patients undergo autologous PBSCT on day 0 per standard of care.
  Interventions: Biological: Anti-CD20 B9E9 scFv-Streptavidin Fusion Protein; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Clearing Agent; Drug: Cytarabine; Drug: Etoposide; Radiation: Indium In 111-DOTA-Biotin; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Pharmacological Study; Radiation: Yttrium Y 90-DOTA-Biotin

INTERVENTIONS:
Biological: Anti-CD20 B9E9 scFv-Streptavidin Fusion Protein — Given IV
  Other Names: Anti-CD20 B9E9 scFv-SA Fusion Protein; Anti-CD20 B9E9-SA Fusion Protein; B9E9 scFvSA Fusion Protein; Recombinant Anti-CD20 B9E9 scFvSA Fusion Protein; scFv B9E9-streptavidin Fusion Protein
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: Autologous Stem Cell Transplantation
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Clearing Agent — Given IV
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Radiation: Indium In 111-DOTA-Biotin — Given IV
  Other Names: In 111-DOTA-Biotin
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Pharmacological Study — Correlative studies
Radiation: Yttrium Y 90-DOTA-Biotin — Given IV
  Other Names: 90Y-DOTA-Biotin; yttrium Y 90 DOTA-biotin

SUMMARY:
This phase I/II trial studies the side effects and best dose of anti-cluster of differentiation (CD)20 radioimmunotherapy (RIT), and to see how well it works when given before chemotherapy and stem cell transplant in treating patients with B-cell malignancies that have not responded to treatment or have come back after responding to treatment. CD20 is a protein found on the cells of a type of cancer cell called B-cells. Anti-CD20 RIT attaches radioactive material to a drug that is designed to target CD20, which brings radioactive material to the cancer cells to kill the cells. This may kill more tumor cells while causing fewer side effects to healthy tissue. Adding anti-CD20 to standard chemotherapy and stem cell transplant may be more effective in treating patients with B-cell malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of 90Y activity that can be delivered via pretargeted radioimmunotherapy (PRIT) using B9E9-fusion protein (B9E9-FP), clearing agent (CA), and radiolabeled tetraazacyclododecane-1,4,7,10-tetraacetic acid (DOTA)-biotin when followed by carmustine, etoposide, cytarabine, and melphalan (BEAM) chemotherapy and autologous stem cell transplantation.

SECONDARY OBJECTIVES:

I. To assess the overall and progression-free survival of the above regimen in such patients.

II. To evaluate the response rates of the above therapy.

III. To evaluate the toxicity and tolerability of the above therapy.

IV. To evaluate the feasibility of delivering sequential high-dose PRIT and chemotherapy.

TERTIARY OBJECTIVES:

I. Assess biodistribution and pharmacokinetics of B9E9-FP and radiolabeled DOTA-Biotin.

II. Assess ability of the clearing agent (CA) to remove excess B9E9-FP from the serum.

III. Evaluate the impact, if any, of circulating rituximab on biodistributions.

OUTLINE: This is a phase I, dose-escalation study of yttrium Y 90 DOTA-biotin followed by a phase II study.

B9E9-FP INFUSION: Patients receive B9E9-fusion protein intravenously (IV) over a minimum of 2 hours on day -17.

CLEARING AGENT INFUSION: Patients receive clearing agent IV over a minimum of 30 minutes on day -15.

RADIOBIOTIN INFUSION: Patients receive indium In 111-DOTA-biotin IV and yttrium Y 90 DOTA-biotin IV over 2-5 minutes on day -14.

BEAM CHEMOTHERAPY: Patients receive BEAM chemotherapy comprising carmustine IV over 3 hours on day -7; etoposide IV over 2 hours twice daily (BID) and cytarabine IV over 4 hours BID on days -6 to -3; and melphalan IV over 30 minutes on day -2.

STEM CELL INFUSION: Patients undergo autologous peripheral blood stem cell transplant (PBSCT) on day 0 per standard of care.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of lymphoma expressing the CD20 antigen and generally must have failed at least one prior standard systemic therapy; the exception will be mantle cell lymphoma (MCL) patients, who may be enrolled while in first complete remission (CR) as well as other select high-risk lymphomas (e.g., Burkitt?s, double hit diffuse large B-cell lymphoma [DLBCL], transformed indolent B-cell non-Hodgkin lymphoma [B-NHL], etc.) in accordance with current transplant standard of care for these patients
* Creatinine (Cr) < 2.0
* Bilirubin < 1.5 mg/dL, with the exception of patients thought to have Gilbert?s syndrome, who may have a total bilirubin above 1.5 mg/dL
* All patients eligible for therapeutic study must have (>= 2 x 10^6 CD34/kg) autologous hematopoietic stem cells harvested and cryopreserved
* Patients must have an expected survival of > 60 days and must be free of major infection
* Patients of childbearing potential must agree to abstinence or the use of effective contraception
* DONOR SELECTION: Not applicable; this protocol employs autologous transplantation, utilizing the patient?s own hematopoietic stem cells obtained from either the peripheral blood or bone marrow

Exclusion Criteria:

* Systemic anti-lymphoma therapy given in the previous 30 days before the scheduled 90Y therapy dose
* Inability to understand or give an informed consent
* Prior radiation > 20 Gy to any critical normal organ (e.g., lung, liver, spinal cord, both kidneys) within 1 year of the treatment date
* Active central nervous system lymphoma
* Other serious medical conditions considered to represent contraindications to bone marrow transplant (BMT) (e.g., abnormally decreased cardiac ejection fraction, diffusion capacity of the lung for carbon monoxide [DLCO] < 50% predicted, patient on supplemental oxygen, acquired immune deficiency syndrome [AIDS], etc.)
* Pregnancy or breast feeding
* Prior bone marrow or stem cell transplant
* Southwest Oncology Group (SWOG) performance status >= 2.0
* Known sensitivity to kanamycin and other aminoglycosides; patients with known hypersensitivity to kanamycin or any other aminoglycoside antibiotic will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-11-17 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (PRIT): B9E9-FP INFUSION: Patients receive B9E9-fusion protein IV over a minimum of 2 hours on day -17.
  CLEARING AGENT INFUSION: Patients receive clearing agent IV over a minimum of 30 minutes on day -15.
  RADIOBIOTIN INFUSION: Patients receive indium In 111-DOTA-biotin IV and yttrium Y 90 DOTA-biotin IV over 2-5 minutes on day -14.
  BEAM CHEMOTHERAPY: Patients receive BEAM chemotherapy comprising carmustine IV over 3 hours on day -7; etoposide IV over 2 hours BID and cytarabine IV over 4 hours BID on days -6 to -3; and melphalan IV over 30 minutes on day -2.
  STEM CELL INFUSION: Patients undergo autologous PBSCT on day 0 per standard of care.
  Anti-CD20 B9E9 scFv-Streptavidin Fusion Protein: Given IV
  Autologous Hematopoietic Stem Cell Transplantation: Undergo autologous PBSCT
Period: Overall Study
Arm/Group | Treatment (PRIT)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (PRIT)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 58 [52 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 3
  White | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Yttrium Y 90 DOTA-biotin Defined as the Dose That is Associated With a True Dose Limiting Toxicity (DLT) Rate of 25%, Where a DLT is Defined as a Therapy-related Grade III or IV Bearman (Transplant) Toxicity
Description: Following the completed observation of the final patient, a two-parameter logistic model will be fit to the data, thereby generating a dose-toxicity curve based on the observed DLT rate at the various dose levels visited. Based on this fitted model, the MTD is estimated to be the dose that is associated with a DLT rate of 25%.
Time Frame: Up to 30 days after transplant
Population: This outcome measure was not done. The starting dose level was level 1 (30 mCi/m2) and in the first stage, up to two patients would be treated at escalating doses in 20 mCi/m2 increments until a DLT was observed. With the 3 participants enrolled, only dose level 5 of 12 was achieved before the study was closed early. The Maximum Tolerated Dose was not determined due to small sample size.
Arm/Group | Treatment (PRIT)
Number analyzed (Participants) | 0

2. Secondary Outcome: Dosimetry of Yttrium Y 90 DOTA-biotin
Description: Assessed using OLINDA dosimetry software. The estimated dose to normal organs and tumor sites will be described based on the tumor to normal organ ratios derived from dosimetry estimates coupled with the absorbed dose to normal organs based on the administered activity of yttrium Y 90 DOTA-biotin.
Time Frame: Up to 7 days after infusion
Population: Absorbed dose in target organs.
Measure: Median (Full Range); unit: cGy/mCi
Arm/Group | Treatment (PRIT)
Number analyzed (Participants) | 3
cGy/mCi
  Liver | 2.5 [1.83 to 2.61]
  Spleen | 3.73 [2.4 to 4.17]
  Lungs | 0.229 [0.194 to 0.477]
  Kidneys | 11.4 [5.57 to 11.9]
  Bone Marrow | 3.75 [1.73 to 5.96]
  Brain | 0.229 [0.194 to 0.477]

3. Secondary Outcome: Incidence of Toxicity, Defined According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Descriptive statistics on the number and percent toxicities will be calculated.
Time Frame: Up to 30 days after transplant
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (PRIT): B9E9-FP INFUSION: Patients receive B9E9-fusion protein IV over a minimum of 2 hours on day -17.
  CLEARING AGENT INFUSION: Patients receive clearing agent IV over a minimum of 30 minutes on day -15.
  RADIOBIOTIN INFUSION: Patients receive indium In 111-DOTA-biotin IV and yttrium Y 90 DOTA-biotin IV over 2-5 minutes on day -14.
  BEAM CHEMOTHERAPY: Patients receive BEAM chemotherapy comprising carmustine IV over 3 hours on day -7; etoposide IV over 2 hours BID and cytarabine IV over 4 hours BID on days -6 to -3; and melphalan IV over 30 minutes on day -2.
  STEM CELL INFUSION: Patients undergo autologous PBSCT on day 0 per standard of care.
  Anti-CD20 B9E9 scFv-Streptavidin Fusion Protein: Given IV
Arm/Group | Treatment (PRIT)
Number analyzed (Participants) | 3
Participants
  Serious Adverse Events | 2
  Other (Not Including Serious) Adverse Events | 2

4. Secondary Outcome: Overall Response Rate
Description: Descriptive statistics on the responses will be calculated.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (PRIT)
Number analyzed (Participants) | 3
Participants
  Participants who achieved a CR | 2
  Participants who achieved a PR | 1

5. Secondary Outcome: Overall Survival
Description: Overall survival will be estimated.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (PRIT)
Number analyzed (Participants) | 3
Participants | 2

6. Secondary Outcome: Progression Free Survival (PFS)
Description: If the true 1-year PFS rate using the proposed approach is 54%, then 24 patients will provide 80% power to detect a statistically significant increased rate of PFS from the fixed rate of 30%, based on a one-sample chi-square test with one-sided significance level of 5%.
Time Frame: 1 year from autologous stem cell transplant
Population: This outcome measure was not done since 24 patients were needed to provide 80% power to detect statistical significance. The sample size of 3 patients is too small to determine the true 1-year PFS rate.
Groups:
- Treatment (PRIT): B9E9-FP INFUSION: Patients receive B9E9-fusion protein IV over a minimum of 2 hours on day -17.
  CLEARING AGENT INFUSION: Patients receive clearing agent IV over a minimum of 30 minutes on day -15.
  RADIOBIOTIN INFUSION: Patients receive indium In 111-DOTA-biotin IV and yttrium Y 90 DOTA-biotin IV over 2-5 minutes on day -14.
  BEAM CHEMOTHERAPY: Patients receive BEAM chemotherapy comprising carmustine IV over 3 hours on day -7; etoposide IV over 2 hours BID and cytarabine IV over 4 hours BID on days -6 to -3; and melphalan IV over 30 minutes on day -2.
Arm/Group | Treatment (PRIT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AEs will be collected from the time of first exposure to an investigational agent through the start of BEAM chemotherapy treatment all SAEs and all grades of adverse events will be captured. From the start of BEAM chemotherapy through day +30 post-transplant non-hematologic adverse events of ≥ grade 3, and all serious adverse events will be captured. Beyond day +30 after transplant/discharge from the transplant service until day +100, only SAEs and grade 4 and 5 toxicities will be collected.
Arm/Group | Treatment (PRIT)
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (PRIT) (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Mucositis, Oral (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (PRIT) (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT02483000/Prot_SAP_000.pdf